CLINICAL TRIAL: NCT04569331
Title: Efficacy of Stimulation of the Efferent Loop Prior to the Closure of the Ileostomy Along With Rehabilitation of the Pelvic Floor After the Closure of the Ileostomy, in the Quality of Life of Patients Who Underwent Anterior Resection of the Rectum(ENESP): Randomized Clinical Trial
Brief Title: Efficacy of Stimulation of the Efferent Loop and Rehabilitation of the Pelvic Floor in the Quality of Life of Patients Who Underwent Anterior Resection of the Rectum (ENESP): Randomized Clinical Trial
Acronym: ENESP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Responsible Party: Principal Investigator, Cristina Vidal, Principal Investigator, Althaia Xarxa Assistencial Universitària de Manresa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CEI 19/26
Record Dates: First submitted 2020-09-16; First posted 2020-09-29 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; ileostomy; quality of life; anterior resection syndrome
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial on the efficacy of efferent loop stimulation prior to ileostomy closure together with pelvic floor rehabilitation after closure of the ileostomy, in the quality of life of patients undergoing anterior rectal resection
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients undergoing anterior rectal resection with protective ileostomy will follow routine clinical practice.
  During hospital admission for ileostomy closure surgery, the stoma therapist reinforces the information on the possibility of anterior resection syndrome (ARS) and hygienic-dietary measures. At the level of the ARS, the patient is informed of the possibility of increased frequency of bowel movements, evacuation dysfunction, such as urgency to defecate or feeling of incomplete emptying. At the level of diet, an astringent diet is recommended during the first week after ileostomy closure to avoid liquid stools. It is also recommended at the level of perineal hygiene to use a cleanser with a pH similar to that of the skin, applying the least possible force on the skin, dry gently after each bowel movement and apply a skin protection product to avoid dermatitis associated with incontinence.
- Stimulation of efferent loop and rehabilitation pelvic floor (Experimental): Stimulation of efferent loop: 3 weeks before the ileostomy closure surgery, efferent loop will be stimulated with 250 ml of water and thickened every 48-hours the first two weeks and once daily the thrid week.
  Rehabilitation of pelvic floor: 3 months after the ileostomy closure surgery, patient will be referred to the pelvic floor unit for pelvic floor rehabilitation.
  Interventions: Procedure: Stimulation of efferent loop; Procedure: Rehabilitation pelvic floor

INTERVENTIONS:
Procedure: Stimulation of efferent loop — Stimulation of efferent loop: 3 weeks before the ileostomy closure surgery, efferent loop will be stimulated with 250 ml of water and thickened.
  This procedure consists of introducing through the light efferent loop ileostomy 250 ml of water with thickener every 48-hours during the first two weeks and once daily the thrid week with a Foley catheter. Patient will be provided with all the material and the procedure sheet for all the stimulation of the efferent loop sessions. This technique will be performed at patient's home until the day before the ostomy patient closure surgery.
  Arms: Stimulation of efferent loop and rehabilitation pelvic floor
Procedure: Rehabilitation pelvic floor — 3 months after the closure of the ileostomy, you will be referred to the pelvic floor rehabilitation unit,where will start 15 individual sessions, 2 days a week (8 weeks of sessions), with reeducation of defecatory habits and hygienic-dietary measures, defecation record where assess stool consistency using the Bristol Scale and number of bowel movements that take place in 24 hours, muscle toning exercises (Exercises Kegel), Biofeedback (BF), rectal balloon work to improve sensitivity and accommodation, reeducation of the expulsive maneuver, and perineal block in situations hyperpressive.
  Arms: Stimulation of efferent loop and rehabilitation pelvic floor

SUMMARY:
Many of the patients operated with sphincter preservation will present an alteration of bowel function and defecation. This dysfunction is variable in its symptoms and severity, and manifests itself in the form of urgency, incontinence and fragmentation of faeces, with repeated, incomplete or difficult evacuations. The set of these symptoms constitutes what is known as anterior resection syndrome (ARS), which can negatively influence the quality of life of the operated patients and constitutes the main objective of the study to be investigated.

From this study, the investigators want to evaluate the efficacy of stimulation of the efferent loop prior to the closure of the ileostomy along with rehabilitation of the pelvic floor after the closure of the ileostomy, in the quality of life of patients who underwent anterior resection of the rectum. A non-pharmacological randomized clinical trial will be conducted, comparing a control group (usual clinical practice), with respect to the experimental group where stimulation of the efferent loop will be performed prior to the closure of the ostomy along with pelvic floor rehabilitation after the closure of the latter. The main dependent variable will be the quality of life evaluated according to the QLQ CR-29 questionnaire, and secondary dependent variables will be evaluated postoperative paralytic ileus and the previous resection syndrome using the LARS scale.

DETAILED DESCRIPTION:
Many of the patients operated with sphincter preservation will present an alteration of bowel function and defecation. This dysfunction is variable in its symptoms and severity, and manifests itself in the form of urgency, incontinence and fragmentation of faeces, with repeated, incomplete or difficult evacuations. The set of these symptoms constitutes what is known as anterior resection syndrome (ARS), which can negatively influence the quality of life of the operated patients and constitutes the main objective of the study to be investigated.

From this study, the investigators want to evaluate the efficacy of stimulation of the efferent loop prior to the closure of the ileostomy along with rehabilitation of the pelvic floor after the closure of the ileostomy, in the quality of life of patients who underwent anterior resection of the rectum. A non-pharmacological randomized clinical trial will be conducted, comparing a control group (usual clinical practice), with respect to the experimental group where stimulation of the efferent loop will be performed prior to the closure of the ostomy along with pelvic floor rehabilitation after the closure of the latter. The main dependent variable will be the quality of life evaluated according to the QLQ CR-29 questionnaire, and secondary dependent variables will be evaluated postoperative paralytic ileus and the previous resection syndrome using the LARS scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing scheduled rectal cancer surgery, carriers of a protective ileostomy with a scheduled surgery date for ileostomy closure
* Patients over 18 years of age
* Patients with absence of cognitive deficit (Pfeiffer: 0-2 errors)
* Patients who agree to participate in the study and sign the informed consent

Exclusion Criteria:

* End ileostomy patients
* Patients with active treatment of Qt or Rt
* Patients with some stoma complication such as mucosal prolapse or peristomal hernia
* Patients with fecal incontinence prior to anterior rectal resection surgery (Wexner scale: greater than 3 points)
* Patients who do not agree to participate in the study
* Patients with cognitive deficit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Quality of life related to health (European Organization for the Research and treatment of Cancer Quality of Life Questionnaire (QLQ-CR29). | 1 month post closure of the ileostomy
  The EORTC QLQ CR-29 questionnaire consists of 29 items (Likert scale), with a response scale for each of them from 1 to 4, with the following structure: 1 = Not at All 2 = A little; 3 = Quite a Bit; 4 = Very much. The QLQ-CR29 has five functional and 18 symptom scales. It contains four subscales (urinary frequency (UF), blood and mucus in stool (BMS), stool frequency (SF), and body image (BI)) and 19 single items (urinary incontinence, dysuria, abdominal pain, buttock pain, bloating, dry mouth, hair loss, taste, anxiety, weight, flatulence, fecal incontinence, sore skin, embarrassment, stoma care problems, sexual interest (men), impotence, sexual interest (women), and dyspareunia). Patients are asked to indicate their symptoms during the past week(s). Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
Quality of life related to health (European Organization for the Research and treatment of Cancer Quality of Life Questionnaire (QLQ-CR29). | 3 month post closure of the ileostomy
  The EORTC QLQ CR-29 questionnaire consists of 29 items (Likert scale), with a response scale for each of them from 1 to 4, with the following structure: 1 = Not at All 2 = A little; 3 = Quite a Bit; 4 = Very much. The QLQ-CR29 has five functional and 18 symptom scales. It contains four subscales (urinary frequency (UF), blood and mucus in stool (BMS), stool frequency (SF), and body image (BI)) and 19 single items (urinary incontinence, dysuria, abdominal pain, buttock pain, bloating, dry mouth, hair loss, taste, anxiety, weight, flatulence, fecal incontinence, sore skin, embarrassment, stoma care problems, sexual interest (men), impotence, sexual interest (women), and dyspareunia). Patients are asked to indicate their symptoms during the past week(s). Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
Quality of life related to health (European Organization for the Research and treatment of Cancer Quality of Life Questionnaire (QLQ-CR29). | 6 month post closure of the ileostomy
  The EORTC QLQ CR-29 questionnaire consists of 29 items (Likert scale), with a response scale for each of them from 1 to 4, with the following structure: 1 = Not at All 2 = A little; 3 = Quite a Bit; 4 = Very much. The QLQ-CR29 has five functional and 18 symptom scales. It contains four subscales (urinary frequency (UF), blood and mucus in stool (BMS), stool frequency (SF), and body image (BI)) and 19 single items (urinary incontinence, dysuria, abdominal pain, buttock pain, bloating, dry mouth, hair loss, taste, anxiety, weight, flatulence, fecal incontinence, sore skin, embarrassment, stoma care problems, sexual interest (men), impotence, sexual interest (women), and dyspareunia). Patients are asked to indicate their symptoms during the past week(s). Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
Quality of life related to health (European Organization for the Research and treatment of Cancer Quality of Life Questionnaire (QLQ-CR29). | 12 month post closure of the ileostomy
  The EORTC QLQ CR-29 questionnaire consists of 29 items (Likert scale), with a response scale for each of them from 1 to 4, with the following structure: 1 = Not at All 2 = A little; 3 = Quite a Bit; 4 = Very much. The QLQ-CR29 has five functional and 18 symptom scales. It contains four subscales (urinary frequency (UF), blood and mucus in stool (BMS), stool frequency (SF), and body image (BI)) and 19 single items (urinary incontinence, dysuria, abdominal pain, buttock pain, bloating, dry mouth, hair loss, taste, anxiety, weight, flatulence, fecal incontinence, sore skin, embarrassment, stoma care problems, sexual interest (men), impotence, sexual interest (women), and dyspareunia). Patients are asked to indicate their symptoms during the past week(s). Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.

SECONDARY OUTCOMES:
Low anterior resection syndrome (LARS) | 1 month post closure of the ileostomy
  Low anterior resection syndrome (LARS) score The LARS questionnaire consists of 5 questions which include: gas incontinence, fluid incontinence, stool frequency, fractionation of defecation and defecation urgency. Each question is scored based on the answer; the total can range from 0 to 42 points. According to the score, the patients are classified into two groups: without LARS, which correspond to scores between 0 and 20 points, and with LARS, which range from 21 to 42 points; Furthermore, this second group is subdivided into mild LARS (21 to 29 points) and severe LARS (30 to 42 points).
Low anterior resection syndrome (LARS) | 3 month post closure of the ileostomy
  Low anterior resection syndrome (LARS) score The LARS questionnaire consists of 5 questions which include: gas incontinence, fluid incontinence, stool frequency, fractionation of defecation and defecation urgency. Each question is scored based on the answer; the total can range from 0 to 42 points. According to the score, the patients are classified into two groups: without LARS, which correspond to scores between 0 and 20 points, and with LARS, which range from 21 to 42 points; Furthermore, this second group is subdivided into mild LARS (21 to 29 points) and severe LARS (30 to 42 points).
Low anterior resection syndrome (LARS) | 6 month post closure of the ileostomy
  Low anterior resection syndrome (LARS) score The LARS questionnaire consists of 5 questions which include: gas incontinence, fluid incontinence, stool frequency, fractionation of defecation and defecation urgency. Each question is scored based on the answer; the total can range from 0 to 42 points. According to the score, the patients are classified into two groups: without LARS, which correspond to scores between 0 and 20 points, and with LARS, which range from 21 to 42 points; Furthermore, this second group is subdivided into mild LARS (21 to 29 points) and severe LARS (30 to 42 points).
Low anterior resection syndrome (LARS) | 12 month post closure of the ileostomy
  Low anterior resection syndrome (LARS) score The LARS questionnaire consists of 5 questions which include: gas incontinence, fluid incontinence, stool frequency, fractionation of defecation and defecation urgency. Each question is scored based on the answer; the total can range from 0 to 42 points. According to the score, the patients are classified into two groups: without LARS, which correspond to scores between 0 and 20 points, and with LARS, which range from 21 to 42 points; Furthermore, this second group is subdivided into mild LARS (21 to 29 points) and severe LARS (30 to 42 points).

OTHER OUTCOMES:
Percentatge of patients with postoperative paralytic ileus | In the first 48 hours postoperatively after the closure of the ileostomy
  Auscultation of intestinal peristaltism and emission of gases and depositions.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Vidal Morral, Principal Investigator — Althaia Xarxa Assitencial Universitària de Manresa
Locations (1):
- Althaia Xarxa Assistencial de Manresa, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No